CLINICAL TRIAL: NCT06361264
Title: Clinical Study of Personalized Chemotherapy for Breast Cancer With Low Doses of Cyclophosphamide, Taking Into Account the Reparative Cycle of Tumor Cells
Brief Title: Clinical Study of Personalized Chemotherapy for Breast Cancer With Low Doses of Cyclophosphamide
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: KARANAHAN (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Karanahan
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Karanahan (Experimental): Reparative cycle of tumor cells is assessed at the preliminary stage in in vitro culture. According to the elaborated regimen, the patient receives 4 intravenous cyclophosphamide injections at the dose of 300 mg/m2 in combination with 4 injections of 1-12 mg of DNAmix administered into prominent tumor nidi and lymph depots. The participant receives from 2 to 6 courses of therapy. The interval between courses is 21 days.
  Interventions: Combination Product: Karanahan

INTERVENTIONS:
Combination Product: Karanahan — During the preparatory stage, a tumor sample from participant is harvested intraoperatively. The primary culture is obtained from this tumor tissue sample. Repair cycle time is estimated, and the day when tumor cells are synchronized at the cell cycle G2/M phase is identified. The schedule of administering cyclophosphamide and DNAmix complex composite preparation is calculated according to the resulting time points. According to the elaborated regimen, the participant receives 4 intravenous cyclophosphamide injections at the dose of 300 mg/m2 in combination with 4 injections of 1-12 mg of DNAmix administered into prominent tumor nidi and lymph depots. The participant receives from 2 to 6 courses of therapy. The interval between courses is 21 days.

SUMMARY:
The goal of this study is to evaluate the safety and clinical efficacy of personalized chemotherapy with low doses of cyclophosphamide administered taking into account the reparative cycle of tumor cells in participants with breast cancer (stage IV or disease progression). The main question it aims to answer is: Does personalized chemotherapy of breast cancer with low doses of cyclophosphamide, taking into account the reparative cycle of tumor cells, lead to a significant reduction in tumor size and improvement in the visual status of controlled tumor foci relative to their initial state? During the preparatory stage, a tumor sample from participant is harvested intraoperatively. The primary culture is obtained from this tumor tissue sample. Repair cycle time is estimated, and the day when tumor cells are synchronized at the cell cycle G2/M phase is identified. The schedule of administering cyclophosphamide and DNAmix complex composite preparation is calculated according to the resulting time points. According to the elaborated regimen, the participant receives 4 intravenous cyclophosphamide injections at the dose of 300 mg/m2 in combination with 4 injections of 1-12 mg of DNAmix administered into prominent tumor nidi and lymph depots. The participant receives from 2 to 6 courses of therapy. The interval between courses is 21 days.

ELIGIBILITY:
Inclusion Criteria:

* stage IV breast cancer or progression of the disease with the presence of foci accessible for biopsy of tumor material;
* complete awareness of the patient about the prognosis of the disease and the proposed treatment;
* the volume of tumor material required for vital assessment of the time parameters of the individual reparative cycle of tumor cells must be at least 4 cm3;
* tumor cells transferred to primary culture must be in a state of proliferative activity.

Exclusion Criteria:

* severe decompensated cardiovascular, respiratory, hepatic, renal failure;
* presence of an acute infectious disease;
* intolerance to cyclophosphamide;
* severe neutropenia - the content of neutrophils is less than 1000 per 1 μl of blood;
* simultaneous participation in another clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The size of tumor foci | 2 months
  Estimation of the size and visual condition of controlled tumor foci relative to their initial state. Tumor response assessment using the Response Evaluation Criteria In Solid Tumors (RECIST 1.1).

SECONDARY OUTCOMES:
The quality of life score | 2 months
  Changes in participants' quality of life during the therapy (score) according to the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30, version 3.0). The scale ranges in score from 0 to 100. Higher score means higher quality of life.
The immunomodulatory effect | 2 months
  The number of CD4+CD25+FoxP3+ regulatory T cells and CD8+CD107a+ T cells is mesuared in participants' blood before therapy and after 2 months using corresponding antibodies. Increase in number of these cells by 14% or more means the development of the adaptive antitumor immune response.

CONTACTS AND LOCATIONS:
Locations (1):
- Karanahan Llc, Novosibirsk, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No